CLINICAL TRIAL: NCT03001843
Title: Does a Ketamine Infusion Decrease Post Operative Narcotic Consumption After Gastric Bypass Surgery?
Brief Title: Ketamine vs Hydromorphone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB201500836 -A
Record Dates: First submitted 2016-12-13; First posted 2016-12-23 (Estimated); Results first posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Laparoscopic Gastric Bypass; Obesity; Pain, Postoperative
MeSH Terms: conditions — Obesity; Pain, Postoperative | interventions — Ketamine; Narcotics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Non-Ketamine (Active Comparator): This group will receive intraoperative narcotics as is usually done for this surgery. This arm will not receive Ketamine.
  Interventions: Drug: Narcotics; Behavioral: pain scale
- Ketamine (Active Comparator): This group will receive an intraoperative infusion of ketamine rather than narcotics to control pain.
  Interventions: Drug: Ketamine; Behavioral: pain scale

INTERVENTIONS:
Drug: Ketamine — Anesthesia of only Ketamine
  Other Names: Ketalar
  Arms: Ketamine
Drug: Narcotics — The narcotic group will receive no ketamine but rather a more standard anesthetic
  Arms: Non-Ketamine
Behavioral: pain scale — 0-10 pain scale. 0 = no pain and 10 = worst pain

SUMMARY:
This study will help to determine if investigators can minimize narcotic use in laparoscopic gastric bypass patients while maintaining adequate pain control. This will allow investigators to minimize the negative side effects of narcotics which is a goal in this population.

DETAILED DESCRIPTION:
The study will be a head to head observational study of patients who have undergone gastric bypass surgery. The methods of intraoperative anesthesiology will be Ketamine or Narcotic. Both are FDA approved methods of delivering anesthesia.

The amount of narcotics a patient receives is part of the medical record post-operatively will be followed from post-anesthesia care unit (PACU) through to discharge. The amount of narcotics needed to control the patient's pain (converted to morphine equivalent units) and pain scores (a hospital standard measure) will be collected for 48 hours for the study, or until discharge, whichever occurs sooner. The conversion to a morphine equivalent unit allows investigators to compare different narcotics the patient may receive in a more standardized way. The results will be analyzed and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Obese patient presenting for laparoscopic gastric bypass between 18 and 65 years of age

Exclusion Criteria:

* Hypersensitivity, allergy, or contraindications to fentanyl, propofol, or ketamine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Smyth, MSN, Principal Investigator — Shands Hospital at the University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-Ketamine | Ketamine
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Ketamine | Ketamine | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants] — Population: Data not collected
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data not collected
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Pain Measured Based on Pain Medication Used on a Scale of 0-10
Description: Used to translate the dose and route of each of the opioids the patient has received over the last 48 hours to a parenteral morphine equivalent using a standard conversion table. SD standard deviation, mg: milligrams, pain measured on a 0-10 scale
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-Ketamine | Ketamine
Number analyzed (Participants) | 27 | 27
units on a scale | 1.3 (2.2) | 0.7 (1.5)

2. Secondary Outcome: Length of Stay (Hours)
Description: Length of stay compared between the 2 groups in hours.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Non-Ketamine | Ketamine
Number analyzed (Participants) | 27 | 27
hours | 43.6 (20.6) | 39.8 (14.5)

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Non-Ketamine | Ketamine
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-02-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT03001843/Prot_002.pdf
  • Informed Consent Form (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT03001843/ICF_003.pdf